CLINICAL TRIAL: NCT02336451
Title: A Phase II, Multi-center, Open-label, Five-arm Study to Evaluate the Efficacy and Safety of Oral Ceritinib Treatment for Patients With ALK-positive Non-small Cell Lung Cancer (NSCLC) Metastatic to the Brain and/or to Leptomeninges
Brief Title: A Phase II Study to Evaluate the Efficacy and Safety of Oral Ceritinib in Patients With ALK-positive NSCLC Metastatic to the Brain and/or to Leptomeninges
Acronym: Ascend-7
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDK378A2205; 2014-000578-20 (EudraCT Number)
Record Dates: First submitted 2015-01-08; First posted 2015-01-13 (Estimated); Results first posted 2020-02-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: ALK-positive Non-small Cell Lung Cancer
Keywords: ALK-positive; NSCLC; non-small cell lung cancer; brain metastasis; metastatic to the brain and/or to leptomeninges; ceritinib; LDK378; NSCLC metastatic to the brain; leptomeninges harboring a confirmed ALK rearrangement
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — ceritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm 1 (PrALKi=Y, PrBRad=Y) (Experimental): Participants with metastases in the brain without evidence of leptomeningeal carcinomatosis (LC), previously treated with radiation to the brain and with prior exposure to an Anaplastic lymphoma kinase inhibitor (ALK-I). Previous treatment with ALK-I other than crizotinib was not allowed in this arm as of protocol amendment 3 and had to present with active brain lesion defined as a lesion free of any local treatment (like stereotactic radiosurgery or whole brain radiation).
  Interventions: Drug: Ceritinib
- Arm 2 (PrALKi=Y, PrBRad=N) (Experimental): Participants with metastases in the brain without evidence of LC, previously untreated with radiation to the brain but with prior exposure to an ALK-I. Previous treatment with ALK-I other than crizotinib was not allowed in this arm 2 as of protocol amendment 3 and had to present with active brain lesion defined as a lesion free of any local treatment (like stereotactic radiosurgery or whole brain radiation).
  Interventions: Drug: Ceritinib
- Arm 3 (PrALKi=N, PrBRad=Y) (Experimental): Participants with metastases in the brain without evidence of LC, previously treated with radiation to the brain but with no prior exposure to an ALK-I. Participants in this arm had to present with active brain lesion defined as a lesion free of any local treatment (like stereotactic radiosurgery or whole brain radiation).
  Interventions: Drug: Ceritinib
- Arm 4 (PrALKi=N, PrBRad=N) (Experimental): Participants with metastases in the brain without evidence of LC, previously untreated with radiation to the brain and with no prior exposure to an ALK-I. Participants in this arm had to present with active brain lesion defined as a lesion free of any local treatment (like stereotactic radiosurgery or whole brain radiation).
  Interventions: Drug: Ceritinib
- Arm 5 (LepDis) (Experimental): Participants had LC with or without evidence of active lesion at the baseline Gadolinium-enhanced brain magnetic resonance imaging (MRI). Previous treatment with ALK-I other than crizotinib was not allowed in this arm as of protocol amendment 3.
  Interventions: Drug: Ceritinib

INTERVENTIONS:
Drug: Ceritinib — LDK378 is a gelatin capsule, administered orally once daily at a dose of 750 mg (five 150 mg capsules) on a continuous dosing schedule on an empty stomach.
  Other Names: LDK378

SUMMARY:
This was a phase II, multi-center, open-label, five-arm study in which the efficacy and safety of oral ceritinib treatment was assessed in patients with NSCLC metastatic to the brain and/or to leptomeninges harboring a confirmed ALK rearrangement, using the FDA approved Vysis ALK Break Apart FISH Probe Kit (Abbott Molecular Inc.) test and scoring algorithm (including positivity criteria). If documentation of ALK rearrangement as described above was not locally available, a test to confirm ALK rearrangement was performed by a Novartis designated central laboratory. Patients waited for the central laboratory result of the ALK rearrangement status before initiating treatment with ceritinib.

DETAILED DESCRIPTION:
Approximately 160 patients diagnosed with ALK-positive metastatic NSCLC (according to the 7th edition of the AJCC [American Joint Committee on Cancer] Cancer Staging Manual) and active lesions in the brain and/or diagnosed with leptomeningeal carcinomatosis were included in the study, approximately 40 patients in Arm 1 and Arm 2, approximately 30 patients in Arms 3 and Arm 4, and approximately 20 patients in Arm 5. Additional patients were enrolled in Arm 4 to achieve approximately 60 patients in Arms 3 and 4 together (i.e. ALKi naïve patients), if enrollment rate in Arm 3 was slow.

* Arm 1 included patients with metastases in the brain without evidence of leptomeningeal carcinomatosis, previously treated with radiation to the brain and with prior exposure to an ALKi.
* Arm 2 included patients with metastases in the brain without evidence of leptomeningeal carcinomatosis, previously untreated with radiation to the brain but with prior exposure to an ALKi.
* Arm 3 included patients with metastases in the brain without evidence of leptomeningeal carcinomatosis, previously treated with radiation to the brain but with no prior exposure to an ALKi.
* Arm 4 included patients with metastases in the brain without evidence of leptomeningeal carcinomatosis, previously untreated with radiation to the brain and with no prior exposure to an ALKi
* Arm 5 included any patients with leptomeningeal carcinomatosis with or without evidence of active lesion at the baseline Gadolinium-enhanced brain MRI.

Note: Previous treatment with ALK inhibitors other than crizotinib was not allowed in Arms 1, 2, and 5.

Ceritinib was administered orally once daily at a dose of 750 mg (five 150 mg capsules) on a continuous dosing schedule. The treatment period started on Cycle 1 Day 1.

Complete tumor assessments including gadolinium enhanced brain MRI was repeated at Week 8 (on Cycle 3 Day 1) and every 8 weeks (i.e. every 2 cycles) thereafter or earlier if clinically indicated. Safety evaluations included (S)AEs, physical examination, vital signs, ECGs, laboratory parameters and WHO performance status. Blood and CSF samples for PK were also collected.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of metastatic NSCLC according to the 7th edition of the AJCC Cancer Staging Manual. In addition, the NSCLC must harbor an ALK rearrangement, as assessed using the FDA approved Vysis ALK Break Apart FISH Probe Kit (Abbott Molecular Inc.) test and scoring algorithm (including positivity criteria). If documentation of ALK rearrangement as described above was not locally available, a test to confirm ALK rearrangement was to be performed by a Novartis designated central laboratory. Patients had to wait for the central laboratory result of the ALK rearrangement status before initiating treatment with ceritinib
* At least one extracranial measurable lesion as defined by RECIST 1.1. A previously irradiated site lesion could only be counted as a target lesion if there was clear sign of progression since the irradiation.
* Patients could or could not have neurological symptoms but must have been able to swallow and retain oral medication.
* Patients had to be neurologically stable within at least 1 week prior to the first dose of study drug.
* Patients could have received prior chemotherapy, crizotinib (other ALK inhibitors were not allowed), biologic therapy or other investigational agents.
* Patients must have recovered from all toxicities related to prior anticancer therapies to grade ≤ 1 (CTCAE v 4.03). Patients with any grade of alopecia were allowed to enter the study.
* Patient had life expectancy ≥ 6 weeks.
* Patient had a WHO performance status 0-2.

Patients in Arm 1 to 4 had to also meet the following inclusion criteria:

- Patients had to have active brain metastases from NSCLC, confirmed by Gadolinium-enhanced MRI without concomitant leptomeningeal carcinomatosis. Dose of steroids had to be stable for 5 days before the baseline brain MRI.

Patients in Arm 5 had to also meet the following inclusion criteria:

- Patients must have been diagnosed with leptomeningeal carcinomatosis.

Exclusion Criteria:

* Patients who needed whole brain radiation to control the brain metastases. Patients were not eligible unless treated brain lesions were progressive or new brain lesions were observed since the post whole brain radiation therapy MRI.
* Planning of any brain local treatment (including but not limited to surgery, stereotactic radiosurgery, whole brain radiation, intrathecal chemotherapy) following the administration of the first dose of study drug.
* Patient with a concurrent malignancy or history of a malignant disease other than NSCLC that had been diagnosed and/or required therapy within the past 3 years. Exceptions to this exclusion included the following: completely resected basal cell and squamous cell skin cancers, and completely resected carcinoma in situ of any type.
* Patient had impairment of GI function or GI disease that could significantly alter the absorption of ceritinib (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, or malabsorption syndrome).
* Patient was receiving unstable or increasing doses of corticosteroids.
* Patient had other severe, acute, or chronic medical conditions including uncontrolled diabetes mellitus or psychiatric conditions or laboratory abnormalities that in the opinion of the investigator could increase the risk associated with study participation, or that could interfere with the interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (52):
- United States (7):
  - USC Kenneth Norris Comprehensive Cancer Center SC-3, Los Angeles, California
  - Stanford Universtiy Medical Center SC-5, Stanford, California
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Dana Farber Cancer Institute SC-12, Boston, Massachusetts
  - The Ohio State University Comprehensive Cancer Center Ohio State University, Columbus, Ohio
  - Southwestern Regional Medical Center, Tulsa, Oklahoma
  - Seattle Cancer Care Alliance, Seattle, Washington
- Novartis Investigative Site, Auckland, Australia
- Novartis Investigative Site, Leuven, Belgium
- Brazil (7):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Natal, Rio Grande do Norte
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, Itajaí, Santa Catarina
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, São Paulo
- Novartis Investigative Site, Toronto, Ontario, Canada
- France (6):
  - Novartis Investigative Site, Marseille, Bouches Du Rhone
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Saint-Herblain Cédex
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Villejuif
- Germany (2):
  - Novartis Investigative Site, Bad Berka
  - Novartis Investigative Site, Cologne
- Novartis Investigative Site, Pokfulam, Hong Kong, Hong Kong
- Italy (11):
  - Novartis Investigative Site, Livorno, LI
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Messina, ME
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Perugia, PG
  - Novartis Investigative Site, Aviano, PN
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Orbassano, TO
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Napoli
- NKI-AVL, Department of Thoracic-Oncology, Amsterdam, Netherlands
- Novartis Investigative Site, Saint Petersburg, Russia
- Novartis Investigative Site, Singapore, Singapore
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (3):
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Taiwan (2):
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Taipei
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Ankara
- United Kingdom (3):
  - Novartis Investigative Site, Sutton, Surrey
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Chow LQM, Barlesi F, Bertino EM, van den Bent MJ, Wakelee HA, Wen PY, Chiu CH, Orlov S, Chiari R, Majem M, McKeage M, Yu CJ, Garrido P, Hurtado FK, Arratia PC, Song Y, Branle F, Shi M, Kim DW. ASCEND-7: Efficacy and Safety of Ceritinib Treatment in Patients with ALK-Positive Non-Small Cell Lung Cancer Metastatic to the Brain and/or Leptomeninges. Clin Cancer Res. 2022 Jun 13;28(12):2506-2516. doi: 10.1158/1078-0432.CCR-21-1838. PMID 35091443

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 156 patients were enrolled and treated with ceritinib. The FAS (N=156) included all patients who received at least one dose of ceritinib with 42, 40, 12, 44 and 18 patients in arms 1 to 5 respectively. The Safety set was identical to full analysis set in this study.
Pre-assignment Details: Approximately 160 patients were planned to be enrolled.
Period: Overall Study
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Started | 42 | 40 | 12 | 44 | 18
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 42 | 40 | 12 | 44 | 18
Not completed — Adverse Event | 1 | 2 | 0 | 6 | 4
Not completed — Death | 6 | 2 | 3 | 6 | 6
Not completed — Physician Decision | 9 | 6 | 7 | 16 | 3
Not completed — Progressive disease | 23 | 26 | 2 | 14 | 4
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0
Not completed — Patient/guardian decision | 2 | 4 | 0 | 2 | 1

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) comprised of all patients who received at least one dose of ceritinib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis) | Total
Number analyzed (Participants) | 42 | 40 | 12 | 44 | 18 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The Full Analysis Set (FAS) comprised of all patients who received at least one dose of ceritinib.
  years | 48.6 (11.37) | 54.5 (12.32) | 50.0 (9.67) | 51.8 (11.21) | 49.9 (11.38) | 51.3 (11.53)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Full Analysis Set (FAS) comprised of all patients who received at least one dose of ceritinib.
  Participants
    Female | 21 | 19 | 6 | 27 | 9 | 82
    Male | 21 | 21 | 6 | 17 | 9 | 74
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 18 | 11 | 7 | 8 | 3 | 47
  Black | 0 | 0 | 0 | 1 | 0 | 1
  Caucasian | 24 | 27 | 4 | 32 | 15 | 102
  Other | 0 | 2 | 1 | 2 | 0 | 5
  Unknown | 0 | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) Per Investigator Assessment
Description: Overall response rate (ORR) is defined as the percentage of participants with a best overall confirmed response of complete response (CR) or partial response (PR) in the whole body as assessed per RECIST 1.1 by the investigator. CR: Disappearance of all non-nodal target and non-target lesions. In addition, all lymph nodes assigned a target or a non-target lesions must be non-pathological in size (< 10 mm short axis), and no new lesion is identified. PR: When all target lesions have disappeared or there is a decrease by at least 30% in the sum of diameter of all target lesions (taking as reference the baseline sum of diameters) is observed & non-target lesions are not in progression or in complete response.
Time Frame: 43 months
Population: The Full Analysis Set (FAS) comprised of all patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 42 | 40 | 12 | 44 | 18
Percentage of participants | 35.7 [21.6 to 52.0] | 30.0 [16.6 to 46.5] | 50.0 [21.1 to 78.9] | 59.1 [43.2 to 73.7] | 16.7 [3.6 to 41.4]

2. Secondary Outcome: Disease Control Rate (DCR) Per Investigator Assessment
Description: DCR: percentage of parts. with best overall response of CR, PR or stable disease (SD) in the whole body, as assessed per RECIST 1.1 by investigator. CR: Disappearance of all non-nodal target and non-target lesions. In addition, all lymph nodes assigned a target or a non-target lesions must be non-pathological in size (< 10 mm short axis), & no new lesion is identified. PR: When all target lesions have disappeared or there is a decrease by at least 30% in the sum of diameter of all target lesions (taking as reference the baseline sum of diameters) is observed and non-target lesions are not in progression or in complete response. SD: Neither sufficient shrinkage in the target lesion to qualify for PR or CR nor an increase in lesions which would qualify for PD & non-target lesions are not in unequivocal progression.
Time Frame: 43 months
Population: The Full Analysis Set (FAS) comprised of all patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 42 | 40 | 12 | 44 | 18
Percentage of participants | 66.7 [50.5 to 80.4] | 82.5 [67.2 to 92.7] | 66.7 [34.9 to 90.1] | 70.5 [54.8 to 83.2] | 66.7 [41.0 to 86.7]

3. Secondary Outcome: Overall Intracranial Response Rate (OIRR) Per Modified RECIST 1.1 Per Investigator Assessment
Description: OIRR was calculated based on response assessments in the brain for patients having measurable brain metastases at baseline. OIRR was defined as the percentage of participants with a best overall confirmed response of CR or PR in the brain as assessed per modified RECIST 1.1. This was applied to the brain only. CR: Disappearance of all non-nodal target & non-target lesions. All lymph nodes assigned a target or a non-target lesions must be non-pathological in size (< 10 mm short axis), & no new lesion is identified. PR: When all target lesions have disappeared or decreased by at least 30% in the sum of diameter of all target lesions (taking as reference the baseline sum of diameters) & non-target lesions are not in progression or in complete response.
Time Frame: 43 months
Population: A subset of FAS (comprised of all patients who received at least one dose of ceritinib) where participants had measurable brain metastases at baseline.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 28 | 29 | 7 | 33 | 8
Percentage of participants | 39.3 [21.5 to 59.4] | 27.6 [12.7 to 47.2] | 28.6 [3.7 to 71.0] | 51.5 [33.5 to 69.2] | 12.5 [0.3 to 52.7]

4. Secondary Outcome: Overall Intracranial Response Rate (OIRR) Per Modified RECIST 1.1 Per Blinded Independent Review Committee (BIRC) Assessment
Description: as for outcome 3
Time Frame: 43 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 30 | 29 | 6 | 34 | 10
Percentage of participants | 33.3 [17.3 to 52.8] | 24.1 [10.3 to 43.5] | 33.3 [4.3 to 77.7] | 58.8 [40.7 to 75.4] | 20.0 [2.5 to 55.6]

5. Secondary Outcome: Intracranial Disease Control Rate (IDCR) Per Modified RECIST 1.1 Per Investigator Assessment at Weeks 8 & 16
Description: IDCR overall: percentage of participants with a best overall response of CR, PR, SD or non-CR/non-PD in the brain, as assessed per modified RECIST 1.1 by the Investigator. This was applied to the brain only. CR: Disappearance of all non-nodal target & non-target lesions. All lymph nodes assigned a target or a non-target lesions must be non-pathological in size (< 10 mm short axis), & no new lesion is identified. PR: When all target lesions have disappeared or there is a decrease by at least 30% in the sum of diameter of all target lesions (taking as reference the baseline sum of diameters) is observed & non-target lesions are not in progression or in complete response. SD: Neither sufficient shrinkage in the target lesion to qualify for PR or CR nor an increase in lesions which would qualify for PD & non-target lesions are not in unequivocal progression.
Time Frame: Week 8 and Week 16
Population: The Full Analysis Set (FAS) comprised of all patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 42 | 40 | 12 | 44 | 18
Percentage of participants
  IDCR at Week 8 | 71.4 [55.4 to 84.3] | 75.0 [58.8 to 87.3] | 58.3 [27.7 to 84.8] | 68.2 [52.4 to 81.4] | 66.7 [41.0 to 86.7]
  IDCR at Week 16 | 59.5 [43.3 to 74.4] | 62.5 [45.8 to 77.3] | 58.3 [27.7 to 84.8] | 65.9 [50.1 to 79.5] | 50.0 [26.0 to 74.0]

6. Secondary Outcome: Intracranial Disease Control Rate (IDCR) Per Modified RECIST 1.1 Per Investigator Assessment - Overall
Description: as for outcome 5
Time Frame: 43 months
Population: The Full Analysis Set (FAS) comprised of all patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 42 | 40 | 12 | 44 | 18
Percentage of participants | 71.4 [55.4 to 84.3] | 85.0 [70.2 to 94.3] | 75.0 [42.8 to 94.5] | 75.0 [59.7 to 86.8] | 66.7 [41.0 to 86.7]

7. Secondary Outcome: Intracranial Disease Control Rate (IDCR) Per Modified RECIST 1.1 Per BIRC Assessment at Weeks 8 & 16
Description: IDCR overall: percentage of participants with a best overall response of CR, PR, SD or non-CR/non-PD in the brain, as assessed per modified RECIST 1.1 by Investigator. This was applied to the brain only. CR: Disappearance of all non-nodal target & non-target lesions. All lymph nodes assigned a target or a non-target lesions must be non-pathological in size (< 10 mm short axis), & no new lesion is identified. PR: When all target lesions have disappeared or there is a decrease by at least 30% in the sum of diameter of all target lesions (taking as reference the baseline sum of diameters) is observed & non-target lesions are not in progression or in complete response. SD: Neither sufficient shrinkage in the target lesion to qualify for PR or CR nor an increase in lesions which would qualify for PD & non-target lesions are not in unequivocal progression.
Time Frame: Week 8 and Week 16
Population: The Full Analysis Set (FAS) comprised of all patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 42 | 40 | 12 | 44 | 18
Percentage of participants
  IDCR at 8 weeks | 76.2 [60.5 to 87.9] | 80.0 [64.4 to 90.9] | 58.3 [27.7 to 84.8] | 68.2 [52.4 to 81.4] | 66.7 [41.0 to 86.7]
  IDCR at 16 weeks | 69.0 [52.9 to 82.4] | 62.5 [45.8 to 77.3] | 58.3 [27.7 to 84.8] | 68.2 [52.4 to 81.4] | 38.9 [17.3 to 64.3]

8. Secondary Outcome: Intracranial Disease Control Rate (IDCR) Per Modified RECIST 1.1 Per BIRC Assessment - Overall
Description: as for outcome 7
Time Frame: 43 months
Population: The Full Analysis Set (FAS) comprised of all patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 42 | 40 | 12 | 44 | 18
Percentage of participants | 73.8 [58.0 to 86.1] | 85.0 [70.2 to 94.3] | 66.7 [34.9 to 90.1] | 75.0 [59.7 to 86.8] | 66.7 [41.0 to 86.7]

9. Secondary Outcome: Time to Intracranial Tumor Response (TTIR) Per Modified RECIST 1.1 Per Investigator Assessment
Description: TTIR was defined as the time from the date of the first dose of ceritinib to the date of the first documented response (CR or PR) in the brain as assessed per modified RECIST 1.1 criteria for patients with measurable brain metastases at baseline. This was applied to the brain only. CR: Disappearance of all non-nodal target and non-target lesions. In addition, all lymph nodes assigned a target or a non-target lesions must be non-pathological in size (< 10 mm short axis), and no new lesion is identified. PR: When all target lesions have disappeared or there is a decrease by at least 30% in the sum of diameter of all target lesions (taking as reference the baseline sum of diameters) is observed & non-target lesions are not in progression or in complete response.
Time Frame: 43 months
Population: A subset of FAS (comprised of all patients who received at least one dose of ceritinib) where participants had measurable brain metastases at baseline and confirmed CR or PR.
Measure: Median (Full Range); unit: months
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 11 | 8 | 2 | 17 | 1
months | 1.87 [1.7 to 7.5] | 1.84 [1.6 to 9.1] | 3.56 [1.8 to 5.3] | 1.77 [1.3 to 7.4] | 1.80 [1.8 to 1.8]

10. Secondary Outcome: Time to Intracranial Tumor Response (TTIR) Per Modified RECIST 1.1 Per BIRC Assessment
Description: as for outcome 9
Time Frame: 43 months
Population: as for outcome 9
Measure: Median (Full Range); unit: months
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 10 | 7 | 2 | 20 | 2
months | 1.91 [1.7 to 5.6] | 1.68 [1.6 to 7.2] | 6.31 [3.5 to 9.1] | 1.81 [1.3 to 9.2] | 1.22 [0.7 to 1.8]

11. Secondary Outcome: Duration of Intracranial Response (DOIR) by Modified RECIST 1.1 Per Investigator Assessment
Description: Defined as the time from the first documented response (PR or CR) in the brain to the date of the first documented disease progression in the brain or death due to any cause, amongst participants with measurable brain metastases at baseline and a confirmed response (PR or CR) in the brain as per modified RECIST 1.1. This was applied to the brain only. CR: Disappearance of all non-nodal target and non-target lesions. In addition, all lymph nodes assigned a target or a non-target lesions must be non-pathological in size (< 10 mm short axis), and no new lesion is identified. PR: When all target lesions have disappeared or there is a decrease by at least 30% in the sum of diameter of all target lesions (taking as reference the baseline sum of diameters) is observed & non-target lesions are not in progression or in complete response.
Time Frame: 43 months
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 11 | 8 | 2 | 17 | 1
months | 9.2 [3.7 to NA] — NA: Not estimable due to small number of responders | 10.1 [3.8 to 17.3] | NA [NA to NA] — NA: Not estimable due to no responders | 7.5 [5.6 to 11.2] | 5.5 [NA to NA] — NA:there was only 1 responder in arm 5, for which the 95% CI was not estimable using Kaplan-Meier method

12. Secondary Outcome: Duration of Intracranial Response (DOIR) by Modified RECIST 1.1 Per BIRC Assessment
Description: Defined as the time from the first documented response (PR or CR) in the brain to the date of the first documented disease progression in the brain or death due to any cause, amongst participants with measurable brain metastases at baseline and a confirmed response (PR or CR) in the brain as per modified RECIST 1.1. CR: Disappearance of all non-nodal target and non-target lesions. In addition, all lymph nodes assigned a target or a non-target lesions must be non-pathological in size (< 10 mm short axis), and no new lesion is identified. PR: When all target lesions have disappeared or there is a decrease by at least 30% in the sum of diameter of all target lesions (taking as reference the baseline sum of diameters) is observed & non-target lesions are not in progression or in complete response.
Time Frame: 43 months
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 10 | 7 | 2 | 20 | 2
months | 11.0 [3.8 to NA] — NA: Not estimable due to small number of responders | 4.6 [3.5 to 20.3] | NA [18.4 to NA] — NA: Not estimable due to small number of responders | 9.2 [5.7 to 11.3] | 3.4 [2.0 to 4.7]

13. Secondary Outcome: Overall Extracranial Response Rate (OERR) Per RECIST 1.1 Per Investigator & BIRC Assessment
Description: OERR was defined as the percentage of participants with a best overall confirmed response of CR or PR outside of the brain, as assessed per RECIST 1.1. CR: Disappearance of all non-nodal target and non-target lesions. In addition, all lymph nodes assigned a target or a non-target lesions must be non-pathological in size (< 10 mm short axis), and no new lesion is identified. PR: When all target lesions have disappeared or there is a decrease by at least 30% in the sum of diameter of all target lesions (taking as reference the baseline sum of diameters) is observed & non-target lesions are not in progression or in complete response.
Time Frame: 43 months
Population: The Full Analysis Set (FAS) comprised of all patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 42 | 40 | 12 | 44 | 18
Percentage of participants
  OERR per Investigator assessment | 31.0 [17.6 to 47.1] | 42.5 [27.0 to 59.1] | 41.7 [15.2 to 72.3] | 61.4 [45.5 to 75.6] | 22.2 [6.4 to 47.6]
  OERR per BIRC assessment | 26.2 [13.9 to 42.0] | 25.0 [12.7 to 41.2] | 50.0 [21.1 to 78.9] | 61.4 [45.5 to 75.6] | 16.7 [3.6 to 41.4]

14. Secondary Outcome: Extracranial Disease Control Rate (EDCR) Per RECIST 1.1 Per Investigator & BIRC Assessment - Overall
Description: EDCR overall was defined as the percentage of participants with a best overall response of CR, PR or SD outside of the brain as assessed per RECIST 1.1. CR: Disappearance of all non-nodal target and non-target lesions. In addition, all lymph nodes assigned a target or a non-target lesions must be non-pathological in size (< 10 mm short axis), & no new lesion is identified. PR: When all target lesions have disappeared or there is a decrease by at least 30% in the sum of diameter of all target lesions (taking as reference the baseline sum of diameters) is observed and non-target lesions are not in progression or in complete response. SD: Neither sufficient shrinkage in the target lesion to qualify for PR or CR nor an increase in lesions which would qualify for PD & non-target lesions are not in unequivocal progression.
Time Frame: 43 months
Population: The Full Analysis Set (FAS) comprised of all patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 42 | 40 | 12 | 44 | 18
Percentage of participants
  EDCR per Investigator assessment | 69.0 [52.9 to 82.4] | 92.5 [79.6 to 98.4] | 66.7 [34.9 to 90.1] | 72.7 [57.2 to 85.0] | 72.2 [46.5 to 90.3]
  EDCR per BIRC assessment | 64.3 [48.0 to 78.4] | 80.0 [64.4 to 90.9] | 66.7 [34.9 to 90.1] | 68.2 [52.4 to 81.4] | 72.2 [46.5 to 90.3]

15. Secondary Outcome: Extracranial Disease Control Rate (EDCR) Per RECIST 1.1 Per Investigator & BIRC Assessment at Weeks 8 & 16
Description: EDCR at weeks 8 & 16: defined as percentage of parts. with CR, PR or SD outside of the brain at Wk 8 & 16 extracranial tumor evaluations respectively, per RECIST 1.1. CR: Disappearance of all non-nodal target and non-target lesions. In addition, all lymph nodes assigned a target or a non-target lesions must be non-pathological in size (< 10 mm short axis), & no new lesion is identified. PR: When all target lesions have disappeared or there is a decrease by at least 30% in the sum of diameter of all target lesions (taking as reference the baseline sum of diameters) is observed and non-target lesions are not in progression or in complete response. SD: Neither sufficient shrinkage in the target lesion to qualify for PR or CR nor an increase in lesions which would qualify for PD & non-target lesions are not in unequivocal progression.
Time Frame: Week 8 and Week 16
Population: The Full Analysis Set (FAS) comprised of all patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 42 | 40 | 12 | 44 | 18
Percentage of participants
  EDCR per Investigator @ Week 8 | 69.0 [52.9 to 82.4] | 82.5 [67.2 to 92.7] | 58.3 [27.7 to 84.8] | 63.6 [47.8 to 77.6] | 72.2 [46.5 to 90.3]
  EDCR per Investigator @ Week 16 | 57.1 [41.0 to 72.3] | 82.5 [67.2 to 92.7] | 66.7 [34.9 to 90.1] | 65.9 [50.1 to 79.5] | 50.0 [26.0 to 74.0]
  EDCR per BIRC @ Week 8 | 66.7 [50.5 to 80.4] | 72.5 [56.1 to 85.4] | 58.3 [27.7 to 84.8] | 61.4 [45.5 to 75.6] | 72.2 [46.5 to 90.3]
  EDCR per BIRC @ Week 16 | 54.8 [38.7 to 70.2] | 70.0 [53.5 to 83.4] | 66.7 [34.9 to 90.1] | 68.2 [52.4 to 81.4] | 44.4 [21.5 to 69.2]

16. Secondary Outcome: Time to Extracranial Tumor Response (TTER) Per RECIST 1.1 Per Investigator Assessment
Description: TTER was defined as the time from the date of the first dose of ceritinib to the date of the first documented response (CR or PR) outside of the brain as assessed per RECIST 1.1 criteria. CR: Disappearance of all non-nodal target and non-target lesions. In addition, all lymph nodes assigned a target or a non-target lesions must be non-pathological in size (< 10 mm short axis), and no new lesion is identified. PR: When all target lesions have disappeared or there is a decrease by at least 30% in the sum of diameter of all target lesions (taking as reference the baseline sum of diameters) is observed & non-target lesions are not in progression or in complete response.
Time Frame: 43 months
Population: A subset of FAS (comprised of all patients who received at least one dose of ceritinib) where participants had confirmed CR or PR.
Measure: Median (Full Range); unit: months
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 13 | 17 | 5 | 27 | 4
months | 1.87 [1.7 to 18.2] | 1.87 [1.6 to 9.3] | 1.81 [1.2 to 12.7] | 1.77 [1.3 to 5.7] | 2.73 [1.8 to 3.6]

17. Secondary Outcome: Time to Extracranial Tumor Response (TTER) Per RECIST 1.1 Per BIRC Assessment
Description: as for outcome 16
Time Frame: 43 months
Population: as for outcome 16
Measure: Median (Full Range); unit: months
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 10 | 6 | 4 | 27 | 4
months | 1.81 [1.7 to 12.9] | 1.86 [1.6 to 22.9] | 2.66 [1.7 to 5.5] | 1.77 [1.3 to 22.0] | 1.81 [1.8 to 1.9]

18. Secondary Outcome: Duration of Extracranial Response (DOER) Per RECIST 1.1 Per Investigator Assessment
Description: DOER was defined as the time from the first documented response (PR or CR) outside of the brain to the date of the first documented disease progression outside of the brain or death due to any cause, amongst patients with a confirmed response (PR or CR) outside of the brain per RECIST 1.1. CR: Disappearance of all non-nodal target and non-target lesions. In addition, all lymph nodes assigned a target or a non-target lesions must be non-pathological in size (< 10 mm short axis), and no new lesion is identified. PR: When all target lesions have disappeared or there is a decrease by at least 30% in the sum of diameter of all target lesions (taking as reference the baseline sum of diameters) is observed & non-target lesions are not in progression or in complete response.
Time Frame: 43 months
Population: as for outcome 16
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 13 | 17 | 5 | 27 | 4
months | 18.4 [5.6 to NA] — NA = Not estimable due to small number of responders | 19.3 [5.7 to NA] — NA = Not estimable due to small number of responders | NA [NA to NA] — NA = Not estimable due to no responders | NA [24.4 to NA] — NA = Not estimable due to small number of responders | 4.6 [1.9 to NA] — NA = Not estimable due to small sample size

19. Secondary Outcome: Duration of Extracranial Response (DOER) Per RECIST 1.1 Per BIRC Assessment
Description: as for outcome 18
Time Frame: 43 months
Population: as for outcome 16
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 11 | 10 | 6 | 27 | 3
months | NA [5.5 to NA] — NA = Not estimable due to small number of responders | 6.0 [3.7 to 27.7] | NA [16.5 to NA] — NA = Not estimable due to small sample size | NA [11.5 to NA] — NA = Not estimable due to small number of responders | 5.5 [3.8 to NA] — NA = Not estimable due to small sample size

20. Secondary Outcome: Overall Response Rate (ORR) (Whole Body) Per RECIST 1.1 Per BIRC Assessment
Description: Overall response rate ORR is defined as the percentage of participants with a best overall confirmed response of complete response (CR) or partial response (PR) in the whole body as assessed per RECIST 1.1 by BIRC. CR: Disappearance of all non-nodal target and non-target lesions. In addition, all lymph nodes assigned a target or a non-target lesions must be non-pathological in size (< 10 mm short axis), and no new lesion is identified. PR: When all target lesions have disappeared or there is a decrease by at least 30% in the sum of diameter of all target lesions (taking as reference the baseline sum of diameters) is observed & non-target lesions are not in progression or in complete response.
Time Frame: 43 months
Population: The Full Analysis Set (FAS) comprised of all patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 42 | 40 | 12 | 44 | 18
Percentage of participants | 23.8 [12.1 to 39.5] | 15.0 [5.7 to 29.8] | 33.3 [9.9 to 65.1] | 61.4 [45.5 to 75.6] | 11.1 [1.4 to 34.7]

21. Secondary Outcome: Disease Control Rate (DCR) (Whole Body) Per RECIST 1.1 Per BIRC Assessment
Description: DCR: defined as percentage of participants with a best overall response of CR, PR or stable disease (SD) in the whole body, per RECIST 1.1 by BIRC. CR: Disappearance of all non-nodal target and non-target lesions. In addition, all lymph nodes assigned a target or a non-target lesions must be non-pathological in size (< 10 mm short axis), & no new lesion is identified. PR: When all target lesions have disappeared or there is a decrease by at least 30% in the sum of diameter of all target lesions (taking as reference the baseline sum of diameters) is observed and non-target lesions are not in progression or in complete response. SD: Neither sufficient shrinkage in the target lesion to qualify for PR or CR nor an increase in lesions which would qualify for PD & non-target lesions are not in unequivocal progression.
Time Frame: 43 months
Population: The Full Analysis Set (FAS) comprised of all patients who received at least one dose of ceritinib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 42 | 40 | 12 | 44 | 18
Percentage of participants | 61.9 [45.6 to 76.4] | 80.0 [64.4 to 90.9] | 66.7 [34.9 to 90.1] | 68.2 [52.4 to 81.4] | 72.2 [46.5 to 90.3]

22. Secondary Outcome: Time to Tumor Response (TTR) (Whole Body) Per RECIST 1.1 Per Investigator Assessment
Description: TTR was defined as the time from the date of the first dose of ceritinib to the date of the first documented response (CR or PR) in the whole body as assessed per RECIST 1.1 criteria per Investigator. CR: Disappearance of all non-nodal target and non-target lesions. In addition, all lymph nodes assigned a target or a non-target lesions must be non-pathological in size (< 10 mm short axis), and no new lesion is identified. PR: When all target lesions have disappeared or there is a decrease by at least 30% in the sum of diameter of all target lesions (taking as reference the baseline sum of diameters) is observed & non-target lesions are not in progression or in complete response.
Time Frame: 43 months
Population: as for outcome 16
Measure: Median (Full Range); unit: months
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 15 | 12 | 6 | 26 | 3
months | 1.87 [1.7 to 9.3] | 2.00 [1.7 to 9.3] | 1.82 [1.2 to 30.1] | 1.81 [1.3 to 3.7] | 1.91 [1.8 to 3.6]

23. Secondary Outcome: Time to Tumor Response (TTR) (Whole Body) Per RECIST 1.1 Per BIRC Assessment
Description: TTR was defined as the time from the date of the first dose of ceritinib to the date of the first documented response (CR or PR) in the whole body as assessed by RECIST 1.1 criteria per BIRC assessment. CR: Disappearance of all non-nodal target and non-target lesions. In addition, all lymph nodes assigned a target or a non-target lesions must be non-pathological in size (< 10 mm short axis), and no new lesion is identified. PR: When all target lesions have disappeared or there is a decrease by at least 30% in the sum of diameter of all target lesions (taking as reference the baseline sum of diameters) is observed & non-target lesions are not in progression or in complete response.
Time Frame: 43 months
Population: as for outcome 16
Measure: Median (Full Range); unit: months
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 10 | 6 | 4 | 27 | 2
months | 2.00 [1.7 to 12.9] | 1.76 [1.6 to 1.9] | 1.82 [1.7 to 26.5] | 1.81 [1.3 to 22.0] | 1.86 [1.8 to 1.9]

24. Secondary Outcome: Duration of Response (DOR) (Whole Body) Per RECIST 1.1 Per Investigator Assessment
Description: DOR was defined as the time from the first documented response (PR or CR) to the date of the first documented disease progression or death due to any cause, amongst patients with a confirmed response (PR or CR) in the whole body per RECIST 1.1 per Investigator. CR: Disappearance of all non-nodal target and non-target lesions. In addition, all lymph nodes assigned a target or a non-target lesions must be non-pathological in size (< 10 mm short axis), and no new lesion is identified. PR: When all target lesions have disappeared or there is a decrease by at least 30% in the sum of diameter of all target lesions (taking as reference the baseline sum of diameters) is observed & non-target lesions are not in progression or in complete response.
Time Frame: 43 months
Population: as for outcome 16
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 15 | 12 | 6 | 26 | 3
months | 10.8 [4.1 to NA] — NA =Not estimable due to small sample size | 12.8 [3.7 to 17.3] | NA [11.7 to NA] — NA = Not estimable due to small number of responders/sample size | 9.2 [7.3 to 23.9] | 5.5 [3.7 to 9.9]

25. Secondary Outcome: Duration of Response (DOR) (Whole Body) Per RECIST 1.1 Per BIRC Assessment
Description: DOR was defined as the time from the first documented response (PR or CR) to the date of the first documented disease progression or death due to any cause, amongst patients with a confirmed response (PR or CR) in the whole body per RECIST 1.1 per BIRC. CR: Disappearance of all non-nodal target and non-target lesions. In addition, all lymph nodes assigned a target or a non-target lesions must be non-pathological in size (< 10 mm short axis), and no new lesion is identified. PR: When all target lesions have disappeared or there is a decrease by at least 30% in the sum of diameter of all target lesions (taking as reference the baseline sum of diameters) is observed & non-target lesions are not in progression or in complete response.
Time Frame: 43 months
Population: as for outcome 16
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 10 | 6 | 4 | 27 | 2
months | 11.0 [2.0 to NA] — NA = Not estimable due to small sample size | 10.6 [3.7 to 20.3] | NA [16.5 to NA] — NA = Not estimable due to small sample size | 9.2 [5.7 to 14.3] | 5.7 [5.5 to 6.0]

26. Secondary Outcome: Progression Free Survival (PFS) (Whole Body) Per RECIST 1.1 Per Investigator & BIRC Assessment
Description: PFS was defined as the time from the date of the first dose of ceritinib to the date of the first radiologically documented disease progression in the whole body per RECIST 1.1 or death due to any cause. A patient who had not progressed or died at the date of the analysis was censored at the time of the last adequate tumor evaluation on or before the cut-off date.
Time Frame: 43 months
Population: The Full Analysis Set (FAS) comprised of all patients who received at least one dose of ceritinib
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 42 | 40 | 12 | 44 | 18
months
  PFS per Investigator assessment: number analyzed (Participants) | 32 | 35 | 6 | 33 | 14
  PFS per Investigator assessment | 7.2 [3.3 to 10.9] | 5.6 [3.6 to 9.2] | NA [1.0 to NA] — NA = Not estimable due to small sample size | 7.9 [5.5 to 9.4] | 5.2 [1.6 to 7.2]
  PFS per BIRC assessment: number analyzed (Participants) | 34 | 36 | 8 | 33 | 14
  PFS per BIRC assessment | 5.0 [3.3 to 9.1] | 5.5 [3.6 to 7.3] | 15.5 [1.0 to NA] — NA = Not estimable due to small sample size | 7.7 [5.5 to 9.7] | 3.6 [1.6 to 5.4]

27. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as time from the date of first dose of ceritinib to the date of death due to any cause. The OS time for patients who were alive at the end of the study or were lost to follow-up was censored at the date of last contact.
Time Frame: 24 weeks
Population: The Full Analysis Set (FAS) comprised of all patients who received at least one dose of ceritinib
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis)
Number analyzed (Participants) | 42 | 40 | 12 | 44 | 18
months | 24.0 [12.6 to NA] — NA = Not estimable due to small number of responders | NA [16.2 to NA] — NA = Not estimable due to small number of responders | NA [1.0 to NA] — NA = Not estimable due to small sample size | NA [26.5 to NA] — NA = Not estimable due to small number of responders | 7.2 [1.6 to 16.9]

28. Secondary Outcome: Pharmacokinetics (PK) of Ceritinib in Study Population: Cmax & Cmin (Trough)
Description: Cmax is the maximum (peak) concentration of drug in plasma. Cmin is the minimum (trough) concentration of drug in plasma. Sparse blood samples for ceritinib PK evaluation in plasma were collected on C1D1 up to C6D1 from all patients who received at least one dose of investigational study treatment.
Time Frame: Cmax: Cycle 2 Day 1 (C2D1); Cmin: C1D1, C1D8, C1D15, C2D1, C3D1, C4D1, C5D1, C6D1 - all 0hr (pre dose)
Population: The Pharmacokinetic Analysis Set (PAS) comprised of all the patients who received at least one (full or partial) dose of ceritinib and provided at least one evaluable PK blood sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Ceritinib 750mg: Participants all received a dose of 750 mg orally in fasted state
Arm/Group | Ceritinib 750mg
Number analyzed (Participants) | 145
ng/mL
  Cmin C1D1: 0hr. (pre dose): number analyzed (Participants) | 130
  Cmin C1D1: 0hr. (pre dose) | 0 (0.0)
  Cmin C1D8: 0hr. (pre dose): number analyzed (Participants) | 107
  Cmin C1D8: 0hr. (pre dose) | 658 (59.2)
  Cmin C1D15: 0hr. (pre dose): number analyzed (Participants) | 106
  Cmin C1D15: 0hr. (pre dose) | 846 (52.9)
  Cmin C2D1: 0hr. (pre dose): number analyzed (Participants) | 84
  Cmin C2D1: 0hr. (pre dose) | 1000 (50.0)
  Cmax C2D1: 4 - 10 hrs. (post dose): number analyzed (Participants) | 73
  Cmax C2D1: 4 - 10 hrs. (post dose) | 1100 (47.8)
  Cmin C3D1: 0hr. (pre dose): number analyzed (Participants) | 61
  Cmin C3D1: 0hr. (pre dose) | 982 (59.1)
  Cmin C4D1: 0hr. (pre dose): number analyzed (Participants) | 46
  Cmin C4D1: 0hr. (pre dose) | 978 (75.4)
  Cmin C5D1: 0hr. (pre dose): number analyzed (Participants) | 45
  Cmin C5D1: 0hr. (pre dose) | 885 (75.5)
  Cmin C6D1: 0hr. (pre dose): number analyzed (Participants) | 40
  Cmin C6D1: 0hr. (pre dose) | 785 (120.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of approx. 168 weeks.
Description: Adverse Event (AE): Any sign or symptom that occurs during the study treatment plus 30 days post treatment.
Groups:
- Arm 4 (PrALKi=N, PrBRad=N): Participants with metastases in the brain without evidence of LC, previously untreated with radiation to the brain and with no prior exposure to an ALK-I. Participants in this arm had to present with active brain lesion defined as a lesion free of any local treatment (like stereotactic radiosurgery or whole brain radiation
- All Participants: All participants who participated in the study and received at least one (full or partial) dose of ceritinib and provided at least one evaluable PK blood sample
Arm/Group | Arm 1 (PrALKi=Y, PrBRad=Y) | Arm 2 (PrALKi=Y, PrBRad=N) | Arm 3 (PrALKi=N, PrBRad=Y) | Arm 4 (PrALKi=N, PrBRad=N) | Arm 5 (LepDis) | All Participants
All-Cause Mortality (participants affected / at risk) | 8/42 | 5/40 | 3/12 | 6/44 | 9/18 | 31/156
Serious Adverse Events (participants affected / at risk) | 28/42 | 17/40 | 4/12 | 15/44 | 11/18 | 75/156
Other Adverse Events (participants affected / at risk) | 42/42 | 40/40 | 11/12 | 43/44 | 18/18 | 154/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (PrALKi=Y, PrBRad=Y) (N=42) | Arm 2 (PrALKi=Y, PrBRad=N) (N=40) | Arm 3 (PrALKi=N, PrBRad=Y) (N=12) | Arm 4 (PrALKi=N, PrBRad=N) (N=44) | Arm 5 (LepDis) (N=18) | All Participants (N=156)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 2 | 0 | 0 | 1 | 0 | 3
Pericarditis (Cardiac disorders) | 2 | 2 | 0 | 0 | 0 | 4
Tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0 | 0 | 2
Keratitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Oesophagopleural fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Disease progression (General disorders) | 0 | 1 | 0 | 0 | 1 | 2
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hyperthermia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 2
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 1 | 3
Sudden death (General disorders) | 1 | 0 | 0 | 1 | 0 | 2
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1
Colonic abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Lung infection pseudomonal (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Nocardia sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 4 | 4 | 1 | 1 | 2 | 12
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
General physical condition abnormal (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Inflammatory marker increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 3 | 1 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 1
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 2
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 2
Dysmetria (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 3
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Memory impairment (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1
Partial seizures (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 3 | 0 | 0 | 2 | 1 | 6
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1
Bradyphrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 2
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 2
Vascular purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Aortic aneurysm rupture (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Embolism (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1 (PrALKi=Y, PrBRad=Y) (N=42) | Arm 2 (PrALKi=Y, PrBRad=N) (N=40) | Arm 3 (PrALKi=N, PrBRad=Y) (N=12) | Arm 4 (PrALKi=N, PrBRad=N) (N=44) | Arm 5 (LepDis) (N=18) | All Participants (N=156)
Anaemia (Blood and lymphatic system disorders) | 8 | 6 | 0 | 5 | 3 | 22
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 2 | 2 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1 | 2
Palpitations (Cardiac disorders) | 1 | 3 | 0 | 0 | 0 | 4
Sinus bradycardia (Cardiac disorders) | 3 | 1 | 0 | 0 | 0 | 4
Vertigo (Ear and labyrinth disorders) | 4 | 0 | 1 | 2 | 0 | 7
Cushingoid (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 1
Vitreous detachment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 5 | 4 | 1 | 1 | 0 | 11
Abdominal pain (Gastrointestinal disorders) | 7 | 12 | 4 | 6 | 4 | 33
Abdominal pain upper (Gastrointestinal disorders) | 6 | 6 | 1 | 10 | 2 | 25
Bowel movement irregularity (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 10 | 9 | 2 | 7 | 4 | 32
Diarrhoea (Gastrointestinal disorders) | 27 | 34 | 8 | 32 | 6 | 107
Dyspepsia (Gastrointestinal disorders) | 7 | 6 | 1 | 2 | 0 | 16
Dysphagia (Gastrointestinal disorders) | 3 | 1 | 1 | 0 | 0 | 5
Epigastric discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 1 | 3
Faecaloma (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Mouth ulceration (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 0 | 5
Nausea (Gastrointestinal disorders) | 23 | 29 | 8 | 19 | 8 | 87
Stomatitis (Gastrointestinal disorders) | 3 | 2 | 0 | 1 | 0 | 6
Vomiting (Gastrointestinal disorders) | 22 | 24 | 4 | 13 | 9 | 72
Asthenia (General disorders) | 11 | 9 | 4 | 9 | 5 | 38
Fatigue (General disorders) | 13 | 14 | 3 | 9 | 3 | 42
Feeling cold (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Gait disturbance (General disorders) | 4 | 0 | 0 | 1 | 1 | 6
General physical health deterioration (General disorders) | 0 | 1 | 1 | 1 | 0 | 3
Hyperthermia (General disorders) | 1 | 0 | 1 | 0 | 0 | 2
Influenza like illness (General disorders) | 2 | 0 | 0 | 3 | 0 | 5
Malaise (General disorders) | 0 | 3 | 1 | 0 | 1 | 5
Non-cardiac chest pain (General disorders) | 9 | 7 | 1 | 3 | 0 | 20
Oedema peripheral (General disorders) | 8 | 6 | 1 | 2 | 2 | 19
Pain (General disorders) | 1 | 0 | 0 | 1 | 2 | 4
Pyrexia (General disorders) | 6 | 14 | 0 | 3 | 1 | 24
Influenza (Infections and infestations) | 1 | 2 | 1 | 2 | 0 | 6
Mucosal infection (Infections and infestations) | 2 | 1 | 0 | 0 | 1 | 4
Nasopharyngitis (Infections and infestations) | 0 | 2 | 1 | 3 | 0 | 6
Oral candidiasis (Infections and infestations) | 2 | 3 | 0 | 1 | 1 | 7
Pneumonia (Infections and infestations) | 1 | 1 | 1 | 0 | 2 | 5
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 2
Tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 2 | 4 | 0 | 11
Urinary tract infection (Infections and infestations) | 3 | 4 | 0 | 2 | 2 | 11
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 18 | 24 | 3 | 23 | 6 | 74
Amylase increased (Investigations) | 2 | 2 | 1 | 3 | 1 | 9
Aspartate aminotransferase increased (Investigations) | 18 | 19 | 2 | 13 | 4 | 56
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 3 | 8 | 1 | 6 | 2 | 20
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blood creatinine increased (Investigations) | 4 | 4 | 2 | 10 | 2 | 22
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 1 | 1
Electrocardiogram QT prolonged (Investigations) | 6 | 1 | 0 | 0 | 1 | 8
Gamma-glutamyltransferase increased (Investigations) | 8 | 13 | 2 | 9 | 3 | 35
Lipase increased (Investigations) | 3 | 0 | 0 | 8 | 2 | 13
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 1 | 0 | 2
Weight decreased (Investigations) | 6 | 8 | 4 | 2 | 3 | 23
Weight increased (Investigations) | 0 | 2 | 0 | 1 | 1 | 4
Decreased appetite (Metabolism and nutrition disorders) | 21 | 14 | 3 | 6 | 6 | 50
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 2 | 1 | 5 | 4 | 16
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 2 | 1 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 2 | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 1 | 0 | 1 | 4 | 14
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 3
Hypophagia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 1 | 0 | 1 | 1 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5 | 2 | 3 | 0 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 8 | 1 | 1 | 0 | 19
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Muscle hypertrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 5 | 0 | 4 | 0 | 12
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 3 | 0 | 0 | 3 | 10
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 2 | 1 | 7
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 1 | 2 | 1 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 2 | 0 | 5
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 1 | 1 | 7
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 2
Aphasia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 2
Balance disorder (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 6 | 8 | 1 | 4 | 3 | 22
Dysarthria (Nervous system disorders) | 1 | 3 | 1 | 1 | 3 | 9
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 5 | 1 | 6
Headache (Nervous system disorders) | 12 | 13 | 3 | 10 | 4 | 42
Memory impairment (Nervous system disorders) | 4 | 1 | 0 | 1 | 1 | 7
Paraesthesia (Nervous system disorders) | 4 | 1 | 0 | 3 | 1 | 9
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Seizure (Nervous system disorders) | 2 | 4 | 0 | 2 | 3 | 11
Somnolence (Nervous system disorders) | 1 | 1 | 0 | 1 | 2 | 5
Tremor (Nervous system disorders) | 1 | 3 | 0 | 1 | 0 | 5
Aggression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Agitation (Psychiatric disorders) | 3 | 0 | 0 | 0 | 1 | 4
Anxiety (Psychiatric disorders) | 1 | 1 | 1 | 1 | 0 | 4
Bradyphrenia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 3 | 0 | 0 | 0 | 0 | 3
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hallucination, auditory (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hallucinations, mixed (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 3 | 4 | 1 | 4 | 1 | 13
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 2
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 8 | 1 | 6 | 4 | 29
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 8 | 2 | 5 | 2 | 21
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 1 | 0 | 4
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 3 | 0 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 1 | 0 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 4 | 1 | 10
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 4 | 0 | 6
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3 | 2 | 1 | 0 | 9
Rash (Skin and subcutaneous tissue disorders) | 4 | 6 | 4 | 7 | 1 | 22
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 2 | 0 | 5
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Skin striae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 3 | 1 | 1 | 1 | 7
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/51/NCT02336451/SAP_000.pdf
  • Study Protocol (2018-05-16): https://cdn.clinicaltrials.gov/large-docs/51/NCT02336451/Prot_001.pdf